CLINICAL TRIAL: NCT06253403
Title: Exploring Sexual Dysfunction in Women Affected by Anorexia Nervosa: Initial Insights
Brief Title: Sexual Dysfunction and Anorexia Nervosa
Acronym: SD&MA
Status: Active, not recruiting | Type: Observational
Sponsor: Comenius University (Other)
Responsible Party: Principal Investigator, Tatiana Hess, Doctoral student, Clinical research, Comenius University
Other Study IDs: study1
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Anorexia Nervosa
Keywords: sexual dysfunction, anorexia nervosa, women, libido
MeSH Terms: conditions — Anorexia Nervosa; Sexual Dysfunction, Physiological | interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- clinic: adult women with anorexia nervosa or actual or after stabilization
  Interventions: Behavioral: psychotherapy
- control: health adult women without any psychological or mental illnes

INTERVENTIONS:
Behavioral: psychotherapy — psychotherapy related to sexual intervention
  Groups: clinic

SUMMARY:
The objective of this observational study is to investigate the potential influence of anorexia nervosa on the sexual health of women. The primary focus is to determine the presence of sexual dysfunction in individuals with anorexia nervosa and explore any potential correlation between eating disorders and sexual dysfunction. To facilitate comparison, data from a control group comprising healthy women is incorporated alongside the clinical group data.

DETAILED DESCRIPTION:
numerous studies indicate that women diagnosed with anorexia nervosa experience a discernible impact on their sexual well-being, often accompanied by symptoms of sexual dysfunction (SD). Such dysfunction may manifest as a diminished libido, reduced sexual desire, and challenges in achieving orgasm

ELIGIBILITY:
Inclusion Criteria:

clinic group :

* adult
* women
* diagnosis of anorexia nervosa
* from Slovakia and Czech Republic

control group:

* health women
* adult
* from Slovakia and Czech Republic

Exclusion Criteria:

clinic group:

* health women
* other diagnosis or disorder
* other country

control group:

* presence of some mental illness
* other country

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects within the clinical group are women diagnosed with either AN or a history of anorexia nervosa
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Female Sexual function index (FSFI) | 1 day
  A self-administered questionnaire was utilized to gather information on participants' sexual experiences and satisfaction over the past four weeks. The questionnaire encompasses six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain, each rated on a scale of 0 to 5. A lower score indicates a higher likelihood of sexual dysfunction.The maximum attainable score is 36 and minimum is 2, with a cut off of 26 serving as a potential diagnostic threshold for sexual dysfunction

SECONDARY OUTCOMES:
The Eating Disorder Examination - Questionnaire Short (EDE-QS | 1 day
  The Eating Disorder Examination - Questionnaire Short (EDE-QS) is a concise 12-item version featuring a 4-point response scale. The maximum attainable score is 36 and minimum is 0, with a cut off of 15 serving as a potential diagnostic threshold for eating disorder. Higher score indicate worse outcome.This instrument is designed to assess eating disorder (ED) symptoms observed within the preceding 7 days. The screening EDE-QS aims to efficiently identify probable ED symptomatology while demonstrating robust psychometric properties.

CONTACTS AND LOCATIONS:
Locations (1):
- Tatiana Hess, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No